CLINICAL TRIAL: NCT07407075
Title: EVALUATION OF THE RELATIONSHIP BETWEEN MUSCLE STRENGTH IMBALANCE AND KINESIOPHOBIA IN POSTOPERATIVE AND CONSERVATIVELY MANAGED MENISCUS PATIENTS
Brief Title: MUSCLE STRENGTH IMBALANCE AND KINESIOPHOBIA IN MENISCUS PATIENTS
Status: Active, not recruiting | Type: Observational
Sponsor: Acıbadem Atunizade Hospital (Other)
Collaborators: Biruni University (Other)
Responsible Party: Principal Investigator, Neslihan Yildizdagi, Pediatric Physiotherapist, Acıbadem Atunizade Hospital
Other Study IDs: Biruni University
Record Dates: First submitted 2026-02-06; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Meniscus Injury; Muscle Strength; Kinesiophobia
Keywords: Meniscus Injuries; Kinesiophobia; BlazePod; Pain
MeSH Terms: conditions — Kinesiophobia; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Post-operative Meniscus Group: This group will consist of individuals who have undergone surgical intervention (meniscectomy or meniscal repair) due to medial meniscal injury confirmed by magnetic resonance imaging (MRI). Participants will be required to have completed at least a three-week postoperative recovery period and to be actively continuing a routine rehabilitation program.
- Conservative Treatment Group: This group will consist of individuals with MRI-confirmed medial meniscal injury who are managed conservatively without surgical intervention and are followed through non-operative approaches such as physiotherapy, exercise, and medical treatment. Participants will be required to have at least two months elapsed since the injury and to be actively engaged in an ongoing rehabilitation program.

SUMMARY:
This study is a cross-sectional and comparative clinical investigation designed to examine the relationship between periarticular muscle strength imbalance and kinesiophobia levels in individuals with meniscal injuries receiving postoperative or conservative treatment, and to determine whether this relationship differs according to the treatment modality.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18 and 50 years of age, with a diagnosis of meniscal injury (male or female)
* Having a medial meniscal injury confirmed by magnetic resonance imaging (MRI)
* Presence of a unilateral injury
* Voluntary agreement to participate in the study
* A minimum of 3 weeks having elapsed since surgery for postoperative participants
* A minimum of 2 months having elapsed since injury for participants receiving conservative treatment

Exclusion Criteria:

* Concomitant anterior cruciate ligament (ACL) injury or additional ligament injuries such as posterior cruciate ligament (PCL), lateral collateral ligament (LCL), or medial collateral ligament (MCL)
* History of fracture or significant trauma to the lower extremity within the past 6 months
* Current or previous neurological disorders (e.g., stroke, multiple sclerosis, peripheral neuropathy, Parkinson's disease)
* Vestibular system disorders or any conditions affecting balance
* Presence of a second surgical intervention or postoperative complications
* Osteoarthritis with a Kellgren-Lawrence grade ≥ 2
* Contracture or severe limitation of knee range of motion restricting joint mobility

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population consists of a total of 50 male and female individuals aged between 18 and 50 years who have been diagnosed with medial meniscal injury and are undergoing either postoperative or conservative treatment.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2026-01-05 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Tampa Kinesiophobia Scale (TKS-17) | Baseline. The evaluation is conducted only once during the research process.
  This is a self-report scale that assesses avoidance of movement and fear of re-injury. It consists of 17 articles. The scale will be completed using a 4-point Likert scale (1=Strongly disagree, 4=Strongly agree), and the total score will range from 17 to 68.
Muscle Strength | Baseline. The assessment will be conducted once during the study period.
  Muscle strength will be assessed using a standardized isometric dynamometer. It will be applied to the quadriceps and hamstring muscles.This will be used to objectively measure isometric muscle strength and determine the difference/asymmetry of strength between the affected and unaffected extremities. This measure quantitatively reflects lower extremity muscle performance and potential functional strength loss.

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) | Baseline. The evaluation will be conducted once during the study period.
  Pain intensity will be assessed using a Visual Analog Scale (VAS) to determine the level of knee pain perceived by participants and will be recorded as a quantitative indicator of subjective pain experience. Pain intensity will be rated on a scale of 0-10. A score of "0" indicates "no pain", and a score of "10" indicates "unbearable pain".
Single Leg Hop Test | Baseline. The evaluation will be conducted once during the study period.
  Functional performance will be assessed using the Single Leg Hop Test, which will provide objective data on the dynamic stability, power generation, and functional capacity of the lower extremity.
International Knee Documentation Committee (IKDC) | Baseline, The evaluation will be conducted once during the study period.
  Participants' knee-related symptoms and functional level will be assessed using the IKDC-SKF. The form consists of items covering symptoms (pain, swelling, locking), activities of daily living, and sports activities, and a score on a scale of 0-100 is obtained; a higher score indicates better function.
Lysholm Knee Scale | Baseline. The evaluation will be conducted once during the study period.
  The Lysholm score is a scale that evaluates knee function on an eight-item scale, scored from 0-100; scores of 92-100 are interpreted as "excellent", 84-91 as "good", 65-83 as "average", and 64 and below as "poor".
Reaction Time Assessment (BlazePod) | Baseline. The evaluation will be conducted once during the study period.
  In this study, the BlazePod Reaction Measurement System will be used to evaluate the neuromuscular response velocity of the lower extremity. The test will last for 60 seconds, the reaction time for each stimulus will be automatically recorded in milliseconds, and the average reaction time will be used in the analysis. A shorter reaction time indicates a better neuromuscular response speed.
Proprioception | Baseline. The evaluation will be conducted once during the study period.
  In this study, the active joint position repetition test will be used to evaluate proprioceptive sensation in the knee joint.

CONTACTS AND LOCATIONS:
Overall Officials: Begüm KARA KAYA, PhD, Principal Investigator — Biruni University
Locations (1):
- Biruni University, Istanbul, Zeytinburnu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available to other researchers due to ethical and confidentiality considerations.